CLINICAL TRIAL: NCT05677269
Title: The (Cost-)Effectiveness of Surgical Excision of Colorectal Endometriosis Compared to ART Treatment Trajectory
Acronym: TOSCA
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Haaglanden Medical Centre (Other); University Medical Center Groningen (Other); Maastricht University Medical Center (Other); Radboud University Medical Center (Other); Reinier de Graaf Groep (Other); Catharina Ziekenhuis Eindhoven (Other); UMC Utrecht (Other)
Responsible Party: Principal Investigator, mdblikkendaal, Principle Investigator, Leiden University Medical Center
Other Study IDs: N22.085
Record Dates: First submitted 2022-12-09; First posted 2023-01-10 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Endometriosis, Rectum; Endometriosis of Colon; Subfertility, Female
Keywords: Colorectal endometriosis; Subfertility; Surgery; In vitro fertilisation; Live birth rate; Quality of life; Cost-effectiveness
MeSH Terms: conditions — Endometriosis; Infertility, Female; Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 40 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colorectal endometriosis patients: Subfertile women between 21 and 40 years with colorectal endometriosis facing the choice between IVF/ICSI or laparoscopic resection of (colorectal) endometriosis.
  Interventions: Procedure: Laparoscopic excision of endometriosis, including colorectal endometriosis; Procedure: In vitro fertilisation or intracytoplasmic sperm injection

INTERVENTIONS:
Procedure: Laparoscopic excision of endometriosis, including colorectal endometriosis — Laparoscopic resection of deep endometriosis, including colorectal endometriosis, in a (candidate) level 2 centre of expertise. Complete resection can exist of either 'shaving' of the nodule from the bowel (leaving the lumen closed), discoid excision or segmental resection, depending on the nodule size and extent of disease.
Procedure: In vitro fertilisation or intracytoplasmic sperm injection — IVF/ICSI treatment trajectory (maximum of 3 cycles), according to the local protocol. Preferably preceded by 3 months downregulation with either Gonadotrophin-releasing hormone (GnRH) analogue or oral contraceptive pill. One IVF/ICSI cycle is defined as the transfer of all the embryos created after one follicle puncture until pregnancy confirmation or failure of the last embryo transfer.

SUMMARY:
To goal of this study is to determine whether laparoscopic resection of colorectal endometriosis results in an increased cumulative live birth rate (CLBR) both spontaneous and after ART (including in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI), and better patient reported outcome measures (PROMs) compared to an IVF/ICSI treatment trajectory.

DETAILED DESCRIPTION:
Endometriosis is characterized by extra-uterine endometrium like tissue and affects 10-15% of the women in their reproductive years and in 5-12% of these women colorectal endometriosis is present. The quality of life is lowered due to severe pain symptoms (dysmenorrhea, dyschezia, dysuria, chronic pelvic pain) and subfertility.The management of colorectal endometriosis-related subfertility is challenging. While the impact of colorectal endometriosis per se remains inconclusive as other intraperitoneal endometriosis lesions are frequently present, fertility is most likely affected by multiple mechanisms including inflammatory alterations in peritoneal fluid, alterations in estrogen and progesterone hormone levels, lowered endometrium receptivity, associated adenomyosis, a lower ovarian reserve (in case endometriomas are present) and adhesion formation that disrupts adnexal anatomy and function. Usually, surgery is preferred in case of dominant pain complaints, while IVF/ICSI is started when the wish to conceive is dominant. Recent evidence suggests a CLBR of 44.9% in patients with rectosigmoid endometriosis treated by surgery compared to 55.9% after 4 cycles of IVF/ICSI treatment without surgery. In the Netherlands, the number of reimbursed IV/ICSI attempts in limited to three. In addition, a combined strategy may result in even higher cumulative live birth rates. However, the place and optimal timing of surgery in patients with colorectal endometriosis and a desire to have children is unknown.

To provide robust evidence that can be extrapolated to the Dutch healthcare system, this study aims to determine whether surgical excision of colorectal endometriosis results in increased CLBR both spontaneous and after IVF/ICSI, and better PROMs compared to an IVF/ICSI treatment trajectory.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal endometriosis defined as endometriosis involving the (colo)rectum:

  #Enzian classification score C1,C2,C3 (C=rectum) or FI (F=far locations, I=sigmoid colon) detected with ultrasound or MRI;
* Women in a heterosexual or in a same-sex relationship;
* The patient has an active wish to conceive and experiences at least one of the following criteria:

  * At least one year of non-conception (either spontaneous of after intra uterine inseminations)
  * Inability to have timed intercourse because of pain (dyspareunia and/or chronic pelvic pain)
  * Severe complaints (expectant management is not acceptable (anymore)
* The patients has an indication for IVF/ICSI according to Dutch guidelines (Werkgroep netwerkrichtlijn, december 2010);

  * failed intra uterine insemination
  * male factor subfertility (oligoasthenoteratozoospermia defined as VCM <1 million)
  * bilateral tubal pathology (e.g. bilateral hydrosalpinx, bilateral tubal occlusion)
  * age > 38 years and (unexplained) subfertility
  * severe endometriosis in case of subfertility
* The patient is faces the choice between IVF/ICSI or laparoscopic (colorectal) endometriosis or is on the waiting list for a respective treatment at T=0 (at the beginning of the treatment trajectory), T=1 (after one unsuccessful IVF/ICSI cycle) or T=2 (after 2 unsuccessful IVF/ICSI cycles)

Exclusion Criteria:

* Patients with deep endometriosis without colorectal involvement;
* Patients who conceive spontaneously prior to intervention;
* Patients requiring surgery on short notice and therefore unable to opt for IVF/ICSI (e.g. in case of unilateral or bilateral hydronephrosis, severe bowel stenosis and suspicion of an impending ileus);
* Patients with a contra-indication for IVF/ICSI (e.g. diminished ovarian reserve (premature ovarian failure) (AMH (when available) <p10 adjusted for age), untreated congenital uterine abnormalities, maltreated/untreated systemic or malignant disease or severe risk factors for oocyte aspiration);
* Patients diagnosed with other diseases causing infertility (e.g. recurrent miscarriages, antiphospholipid syndrome);
* Not able to read and understand Dutch or English.

Ages: 21 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Endometriosis only affects women
Study Population: Subfertile women between 21 and 40 years with colorectal endometriosis facing the choice (at the start of their treatment trajectory or after one or two unsuccessful IVF/ICSI cycles) between IVF/ICSI or laparoscopic excision of (colorectal) endometriosis to increase the chance to conceive (naturally)
Sampling Method: Non-Probability Sample
Enrollment: 339 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative live birth rate | At the end of the study period (live birth or after 3 IVF/ICSI attempts and/or surgery in the follow-up period (40 months) )
  Live birth is defined as the complete expulsion or extraction from a women of a product of fertilization, after 20 weeks of gestational age; which, after such separation, breathes or shows any other evidence of life, such as heart beat, umbilical cord pulsation or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut of the placenta is attached. A birth weight of 350 grams or more can be used if gestational age is unknown

SECONDARY OUTCOMES:
Endometriosis specific symptoms | At baseline (T=0: when informed consent is granted), 12, 24 and 36 months and in case of surgery, before surgery.
  Endometriosis Health Profile-30 (EHP-30). The overall EHP-30 score ranges from 0 to 100, with a high score indicating poorer health-related quality of life.
Quality of life in general | At baseline (T=0: when informed consent is granted), 6, 12, 18, 24, 30, 36 and 40 months and in case of surgery, before surgery.
  EuroQql five-dimensional 5 levels (EQ-5D-5L) and EuroQql Visual Analog Scale (EQ-VAS).
  According to the Dutch scoring algorithm, the EQ-5D-5L score index value ranges from -0.446 (55555 worst health state) to 1 (11111, best health state).
  Overall health will be represented by the EQ-VAS, ranging from 0 to 100, with higher scores indicating better health.
Bowel specific symptoms | At baseline (T=0: when informed consent is granted), 12, 24 and 36 months and in case of surgery, before surgery.
  Lower Anterior Resection Syndrome score (LARS score). The total LARS score ranges from 0, indicating no LARS to 42 points, indicating major LARS.
Pain scores | At baseline (T=0: when informed consent is granted), 12, 24 and 36 months and in case of surgery, before surgery.
  NRS score for dysmenorrhea, dysuria, dyschezia, dyspareunia and chronic pelvic pain. The NRS scale ranges from 0 (no pain) to 10 (worst pain imaginable).
Productivity costs | At baseline (T=6, 12, 18, 24, 30, 36 and 40 months and in case of surgery, before surgery.
  Productivity costs questionnaire: institute for Medical Technology Assessment (iMTA) Productivity Cost Questionnaire (iPCQ).
  Productivity costs will be measured by calculating absence from paid work (absenteeism), reduced productivity at paid work (presenteeism), and productivity loss in unpaid work. Hours of productivity loss will be translated by a standard cost price of productivity per hour.
Medical costs per group | At the end of the study period (live birth or after 3 IVF/ICSI attempts and/or surgery in the follow-up period (40 months) )
  Costs surgery, costs IVF/ICSI treatment, costs extra hospital admissions / emergency room visits / visits outpatient care
Complications | At the end of the study period (live birth or after 3 IVF/ICSI attempts and/or surgery in the follow-up period (40 months) )
  Intraoperative and postoperative complications, IVF/ICSI associated complications, pregnancy complications

CONTACTS AND LOCATIONS:
Overall Officials: Mathijs D. Blikkendaal, MD, PhD, Principal Investigator — Nederlandse Endometriose Kliniek (NEK), Reinier de Graaf Gasthuis; Andries RH Twijnstra, MD, PhD, Study Chair — Leiden University Medical Center; Astrid EP Cantineau, MD, PhD, Study Chair — University Medical Center Groningen; Jacques Maas, MD, PhD, Study Chair — Maastricht University Medical Center; Annemiek Nap, MD, PhD, Study Chair — Radboud University Medical Center; Dana Huppelschoten, Study Chair — Catharina Ziekenhuis; Simone Broer, Study Chair — UMC Utrecht; Tobias Limperg, Study Chair — Nederlandse Endometriose Kliniek (NEK), Reinier de Graaf Gasthuis; Yvonne Louwers, Study Chair — Erasmus Medical Center; Marieke Verberg, Study Chair — Medisch Spectrum Twente
Locations (10):
- Netherlands (10):
  - Catharina Ziekenhuis, Eindhoven
  - Medical Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
  - Radboud university medical center, Nijmegen
  - Erasmus Medical Centre, Rotterdam
  - Haaglanden Medical Center, The Hague
  - Utrecht Medical Center, Utrecht
  - Nederlandse Endometriose Kliniek (Reinier de Graaf Gasthuis), Voorburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] F Barra, C Scala, S Bogliolo, N Di Donato, M Ceccaroni, S Ferrero, O-309 Surgery versus IVF/ICSI in infertile women with rectosigmoid endometriosis: the FERTILITY-RECTOSIGMOID study, Human Reproduction, Volume 37, Issue Supplement_1, July 2022